CLINICAL TRIAL: NCT02186444
Title: Navigator Guided e-Psychoeducational Intervention for Prostate Cancer Patients and Their Caregivers
Brief Title: Navigator Guided e-Psychoeducational Intervention
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-17455
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: newly diagnosed prostate cancer; prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHI Navigator: Personalized Health Information Navigator (PHIN).
  Interventions: Other: Personalized Health Information Navigator (PHIN)
- NCI Information Booklets (IB): National Cancer Institute (NCI) Information Booklets (IB).
  Interventions: Other: NCI Information Booklets (IB)

INTERVENTIONS:
Other: Personalized Health Information Navigator (PHIN) — The application (or "app") titled Personalized Health Information Navigator (PHIN) is an interactive psycho-educational intervention that will be delivered via mobile tablet technology. The PHIN provides patient-centered education. At the first meeting, the community navigator will provide a visual demonstration of PHIN on the Apple iPad. The community navigator will leave the iPad with the participant for 6-weeks and will stress the importance of using the PHIN app to address any educational or psychosocial needs.
  Groups: PHI Navigator
Other: NCI Information Booklets (IB) — Participants will receive a packet of information booklets ("What You Need to Know About Prostate Cancer"; "Taking Time: Support for People with Cancer"; and "Facing Forward, Life After Cancer Treatment") that address prostate cancer treatment options, the late and long term effects, follow-up care, and sources of support. At the first meeting, the community navigator will provide a review of the print materials and stress the importance of reading the booklets carefully to help prepare for the discussion with your healthcare provider. The community navigator will leave the print materials with the participant for 6-weeks.
  Groups: NCI Information Booklets (IB)

SUMMARY:
The purpose of this study is to evaluate the impact of providing newly diagnosed prostate cancer patients and their caregivers with an interactive mobile tablet technology-based application delivered by a community navigator versus providing National Cancer Institute (NCI) information booklets delivered by a Community Navigator (CN) on patient outcomes (decisional satisfaction, quality of life, knowledge, decisional conflict) and shared decision making practices (decision making involvement).

ELIGIBILITY:
Inclusion Criteria:

* Men newly diagnosed (within 6 months) with biopsy confirmed case of prostate cancer
* 40 - 80 years of age
* Able to speak and read English
* Live within 120 miles of a healthcare treatment facility
* Have no documented or observable visual, auditory, psychiatric, or neurological disorders that would interfere with study participation
* Be able to complete telephone interviews
* Have not completed the first course of treatment
* Have a family member/caregiver willing to participate
* Capable of providing written consent for study participation. Men diagnosed with early stage, locally advanced or metastatic disease or men who are on active surveillance will be eligible to participate in this study.
* Caregiver must be aged 18 or older
* Caregiver must be identified by patient as their caregiver (i.e., provider of emotional and/or physical care)
* Caregiver must have not been diagnosed with cancer in the previous year or be receiving cancer treatment

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Moffitt Cancer Center Genitourinary Clinic, University of South Florida Genitourinary Clinic, or community-based urologists and primary care providers.
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Final Survey Results per Study Arm | 6 months post baseline survey
  Investigators plan to assess if the psycho-educational intervention, PHIN, delivered by a CN is more efficacious as compared to NCI Information Booklets (IB) delivered by a CN. Participants will be asked to complete a baseline set of surveys and follow-up surveys at three additional time points: (1) 6 weeks after receiving the educational intervention; (2) after the follow-up decision with their doctor or health care provider; and (3) 6 months after the baseline surveys were done.

CONTACTS AND LOCATIONS:
Overall Officials: B. Lee Green, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer and Research Institute, Tampa, Florida, United States